CLINICAL TRIAL: NCT01509391
Title: Keyhole Limpet Hemocyanin in Chronic Hepatitis C and Compensated Cirrhosis - Pilot Study IM1
Brief Title: Keyhole Limpet Hemocyanin in Chronic Hepatitis C
Acronym: IM1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Rudolf Stauber, MD, Univ. Prof. Dr., Medical University of Graz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCVGRZ-IM1
Record Dates: First submitted 2012-01-09; First posted 2012-01-13 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2012-10

CONDITIONS: Chronic Hepatitis C; Liver Cirrhosis
MeSH Terms: conditions — Hepatitis C, Chronic; Liver Cirrhosis | interventions — keyhole-limpet hemocyanin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Keyhole-limpet hemocyanine (Experimental)
  Interventions: Drug: keyhole-limpet hemocyanin

INTERVENTIONS:
Drug: keyhole-limpet hemocyanin — Subcutaneous administration keyhole-limpet hemocyanin

SUMMARY:
In this study the investigators examine the safety and efficacy of Keyhole-limpet-hemocyanin in patients with chronic hepatitis c infection and liver cirrhosis. The investigators hypothesize that administration of keyhole-limpet-hemocyanin reduces the viral load in patients infected with hepatitis c.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Hepatitis C infection
* no previous therapy
* at least one contraindication to interferon therapy
* liver cirrhosis
* age between 18-80 y
* women of not childbearing age

Exclusion Criteria:

* Hypersensitivity against keyhole-limpet hemocyanin
* previous treatment against hepatitis c
* autoimmune disorders
* immunosuppression
* hepatocellular carcinoma or other malignancies
* coinfection with hepatitis b or HIV
* pregnancy
* cardiovascular event during the last 6 months (stroke or MCI)
* uncontrolled diabetes
* renal insufficiency (GFR < 50 ml/min) or chronic hemodialysis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Hepatitis C viral load at week 24 | 24 weeks

SECONDARY OUTCOMES:
Hepatitis c viral load at weeks 1,2,4,8,12,18,32 | 1,2,4,8,12,18,32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf E Stauber, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria